CLINICAL TRIAL: NCT00842803
Title: Post-Operative Use of Salt Poor Albumin Solution in Resuscitation of Orthotopic Liver Transplant Recipients Status 1-2. A Prospective Randomized Controlled Trial.
Brief Title: Post-Operative Use of Salt Poor Albumin Solution in Resuscitation of Orthotopic Liver Transplant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Dr Peter Metrakos, MUHC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SDR-08-030
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Liver Transplantation
Keywords: Liver; transplant; albumin; outcome; Liver transplant recipients canadian transplant status 1 or 2
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (No Intervention): Patients in this group will not be allowed albumin or any other colloids fluid for the first 7 days post-operative
- Albumin group (Experimental): Patients in this arm will receive albumin infusions 3 times a day for the first 7 days post-operative
  Interventions: Drug: Albumin infusion (25% albumin)

INTERVENTIONS:
Drug: Albumin infusion (25% albumin) — Patients in this arm will receive albumin infusions 3 times a day for the first 7 days post-operative
  Arms: Albumin group

SUMMARY:
The purpose of the study is to examine if outcome after liver transplantation is improved by using albumin infusion post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Canadian Transplant status 1 or 2
* Patients at the Royal Victoria Hospital, Montreal, Canada

Exclusion Criteria:

* Emergency liver transplant (canadian transplant status 3 or 4)
* patients who have received more than 300cc of albumin within 48 hours prior to transplant
* patients who underwent previous solid organ transplant
* multi-organs transplant recipients
* patients who had previous adverse reaction to human albumin solution
* patients who have religious restriction to receiving human blood products.
* patients or surrogate unable to give consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Post Transplant Liver Function Test (PTLFT) | Post-operative Day1 through 7 and Day 15,30, 45

SECONDARY OUTCOMES:
Functional 6 minutes walking test | Post-operative
Calculated creatinine clearance | Post-operative day 1, 7, 15, 30, 45
Length of hospital stay | post-operative
ICU length of stay | post-operative
duration of mechanical ventilation | post-operative
duration of renal replacement therapy | postoperative
ICU readmission rate | post-operative
reintubation rate | post-operative
Post-operative infection rate | Post-operative
Need to re-operation unrelated to technical complication | post-operative
Functional hand grip Jamar Dynamometer hand grip test | Post-op day 7, 15, 30

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada